CLINICAL TRIAL: NCT01264952
Title: Treatment of Liver Metastases With Electrochemotherapy
Acronym: ECTJ
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Collaborators: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-Z 16/KSOPKR-6
Record Dates: First submitted 2010-12-15; First posted 2010-12-22 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Liver Metastases
Keywords: Liver metastases of colorectal cancer; Bleomycin; Electrochemotherapy
MeSH Terms: interventions — Electrochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Electrochemotherapy — Treatment procedure: anesthesia, positioning of electrodes, intravenous in bolus administration of bleomycin (15 mg/m2), within 5-30 min after administration of bleomycin application of electric pulses (8 pulses, duration 100 microseconds, frequency 4 Hz with amplitude adequate to cover the whole treated lesion with electric field necessary for reversible plasma membrane permeabilization), removal of electrodes.
  The maximum duration of procedure is 90 minutes.
  Other Names: Device: Cliniporator Vitae®; Drug: Bleomicin PHC 15 e. (United States Pharmacopeia - USP)

SUMMARY:
The aim of the study is to evaluate toxicity and effectiveness of electrochemotherapy with bleomycin in treatment of liver metastases of colorectal cancer in clinical study phase I and II.

The study will include 10-15 patients with colorectal cancer with synchronous or metachronous liver metastases, but electrochemotherapy will be performed on metastasis not more than 3 cm in the largest diameter.

Treatment effectiveness will be evaluated by magnetic resonance imaging (MRI) and ultrasonography (US) in a monthly interval. Two or three month after the first operation the treated and untreated metastases will be resected and through histological analyses performed.

The secondary objectives of the trial are to quantify the impact of the treatment on the patient's quality of life, tolerance to the therapy and suitability for larger study to be conducted.

DETAILED DESCRIPTION:
The study will be conducted on patients with colorectal cancer with synchronous or metachronous liver metastases. Included will be 10-15 patients.

Predominantly, patients with synchronous metastases will be included into the study. These patients present liver metastases at the time of primary tumor resection. Electrochemotherapy will be performed on one metastasis not more than 3 cm in largest diameter at the time of the primary tumor operation, but patients have to have at least 2 to 8 metastases. These metastases will be aimed to be resected in the following operation. It is a standard procedure that liver metastases are resected 2-3 months after the primary tumor resection, in the meantime they are on standard chemotherapeutic protocol (FOLFOX, FOLFIRI, Capecitabine). Only in the case of solitary metastasis smaller than 3 cm in diameter, it is resected during the resection of the primary tumor. In the study additional antitumor effectiveness of electrochemotherapy to other treatment (chemotherapy) will be evaluated, compared to non-electrochemotherapy treated metastases. Treatment effectiveness will be evaluated by magnetic resonance imaging (MRI) and ultrasonography (US), in a monthly interval. Two to three month after the first operation the treated and untreated metastases will be resected and thorough histological analysis performed.

The second group of patients will be with metachronous liver metastases not larger than 3 cm in diameter, that location is in the vicinity of hollow liver structures and would not be possible to resect them without extensive and potentially jeopardizing liver resection. One of them will be treated by electrochemotherapy. In a month interval treatment effectiveness will be evaluated by MRI. In the case that metastases will decrease in size and to the situation that metastases are resectable, second operation will be performed, metastases resected and thorough histopathological evaluation performed. Otherwise standard treatment procedure will be performed (chemotherapy).

All patients will be treated after the procedure is thoroughly described to them, and have signed informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable liver metastases, presented simultaneously with primary tumor, aimed at primary tumor resection and in a 2-3 month interval resection of liver metastases. One metastasis will be treated by electrochemotherapy, not larger than 3 cm in diameter.
* Metastasis has to be accessible for application of electrochemotherapy during the operation, without major liver manipulation or mobilization in order not to create situation that would hamper feasibility of the second operation; resection of metastases.
* Patients with metachronous liver metastases, that are positioned in unresectable liver area, near blood vessels, but inoperable patients.
* Recurrent liver metastases, not more than 3, that are not larger than 3 cm in diameter.
* Histologically and cytologically confirmed cancer, any histological differentiation.
* Life expectancy more than 3 month.
* Performance status Karnofsky ≥ 70 or (World Health Organization) WHO ≥ 2.
* Age more than 18.
* The patient must be offered standard treatment.
* Electrochemotherapy is offered to the patients in the case of the disease progression during the standard treatment, in the case or metastases recurrence, or when they refuse standard treatment.
* Treatment free interval 2-5 weeks, depending on the drugs used.
* Patient must be mentally capable of understanding the information given.
* Patient must give informed consent.

Exclusion Criteria:

* Metastases more than 3 cm in diameter.
* Synchronous unresectable metastases.
* Metachronous unresectable metastases or bigger than 3 cm in diameter.
* Visceral, bone or diffuse metastases.
* Coagulation disturbances.
* Allergic reaction to bleomycin, or cumulative dose of 250 mg/m2 bleomycin received.
* Impaired kidney function (creatinin > 150 µmol/l).
* Patients with hearth failure or pace maker.
* Patients with epilepsy.
* Secondary primary tumor, except surgically treated noninvasive cancer of cervix, or surgically or irradiated basal cell carcinoma.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-11; Primary Completion 2013-03 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eldar Gadzijev, MD, PhD, Principal Investigator — Institute of Oncology Ljubljana, Department of Surgical Oncology, Ljubljana, Slovenia; Gregor Sersa, PhD (Biol.), Study Director — Institute of Oncology Ljubljana, Department of Experimental Oncology, Ljubljana, Slovenia
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Edhemovic I, Gadzijev EM, Brecelj E, Miklavcic D, Kos B, Zupanic A, Mali B, Jarm T, Pavliha D, Marcan M, Gasljevic G, Gorjup V, Music M, Vavpotic TP, Cemazar M, Snoj M, Sersa G. Electrochemotherapy: a new technological approach in treatment of metastases in the liver. Technol Cancer Res Treat. 2011 Oct;10(5):475-85. doi: 10.7785/tcrt.2012.500224. PMID 21895032

RESULTS

PARTICIPANT FLOW:
Groups:
- Bilateral, Multiple, Metachronous Metastases: The first group included patients with bilateral, multiple, metachronous metastases in whom standard treatment included twostage liver resection, due to the extent of the disease and/or their general condition. During the first operation, right portal vein was ligated and metastases on the left side were excised or ablated with radiofrequency ablation. At the same time, up to three metastases on the right side were treated with electrochemotherapy. During the second operation, both treated and non-treated metastases on the right side were removed with right hemihepatectomy.
- Synchronous Metastases: The second group (group II) included patients with synchronous metastases, but their general condition and extent of the disease did not allow simultaneous removal of the primary tumor and metastases. During the first operation, the primary tumor was removed (colorectal resection) and some of the liver metastases were treated by electrochemotherapy. About 6 weeks later, during the second operation for liver metastases, both treated and non-treated metastases were removed with liver resection.
- <= 3 Metachronous, Unresectable Liver Metastases: The third group included patients with up to three metachronous, unresectable liver metastases, demanding too excessive resection, or untreatable by standard thermal ablative methods, due to the close proximity of major blood vessels. Electrochemotherapy was offered to these patients as the only treatment option.
Period: Overall Study
Arm/Group | Bilateral, Multiple, Metachronous Metastases | Synchronous Metastases | <= 3 Metachronous, Unresectable Liver Metastases
Started | 6 | 2 | 8
Completed | 6 | 2 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group I: Patients with bilateral, multiple, metachronous metastases in whom standard treatment included twostage liver resection, due to the extent of the disease and/or their general condition. During the first operation, right portal vein was ligated and metastases on the left side were excised or ablated with radiofrequency ablation. At the same time, up to three metastases on the right side were treated with electrochemotherapy. During the second operation, both treated and non-treated metastases on the right side were removed with right hemihepatectomy.
- Group II: Patients with synchronous metastases, but their general condition and extent of the disease did not allow simultaneous removal of the primary tumor and metastases. During the first operation, the primary tumor was removed (colorectal resection) and some of the liver metastases were treated by electrochemotherapy. About 6 weeks later, during the second operation for liver metastases, both treated and non-treated metastases were removed with liver resection.
- Group III: Patients with up to three metachronous, unresectable liver metastases, demanding too excessive resection, or untreatable by standard thermal ablative methods, due to the close proximity of major blood vessels. Electrochemotherapy was offered to these patients as the only treatment option.
- Total: Total of all reporting groups
Arm/Group | Group I | Group II | Group III | Total
Number analyzed (Participants) | 6 | 2 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 7 | 12
  >=65 years | 3 | 0 | 1 | 4
Age, Continuous [Median (Standard Deviation); unit: years] | 60.0 (6.4) | 45.5 (19.1) | 57.3 (10.7) | 56.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 4
  Male | 5 | 2 | 5 | 12
Region of Enrollment [Number; unit: participants]
  Slovenia | 6 | 2 | 8 | 16

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Non-Serious Adverse Events
Time Frame: After operation on tha days 2, 7, 30, monthly
Measure: Number; unit: patients with non-severe adverse events
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 6 | 2 | 8
patients with non-severe adverse events | 3 | 2 | 7

2. Secondary Outcome: Treatment Evaluation of Tumor Response - Measurements of Tumor Lesions by Contrast Enhanced Ultrasonography (US-Doppler), Magnetic Resonance Imaging (MRI), Computed Tomography (CT), Histology
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI:
  Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: After operation or 1st day after operation, 7th day, 30th day, monthly
Measure: Number; unit: metastases
Units Other Than Participants: metastases
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 6 | 1 | 8
Number analyzed (metastases) | 12 | 1 | 14
metastases | 10 | 1 | 10

3. Primary Outcome: Evaluation of Toxicity Related to Electrochemotherapy (Toxicity, Symptoms)
Time Frame: After operation on day 7
Measure: Number; unit: events
Arm/Group | Group I | Group II | Group III
Number analyzed (Participants) | 6 | 2 | 8
events | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group I | Group II | Group III
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/2 | 3/8
Other Adverse Events (participants affected / at risk) | 3/6 | 2/2 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I (N=6) | Group II (N=2) | Group III (N=8)
Small bowl obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Colon perforation (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal abcess (Gastrointestinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I (N=6) | Group II (N=2) | Group III (N=8)
Infection NOS (Infections and infestations) | 3 | 1 | 6
Fever (Infections and infestations) | 2 | 0 | 0
Atrial fibrilation (Cardiac disorders) | 1 | 0 | 0
Pulmonary hypertension (Vascular disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Wound infection (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Transient liver failure (Hepatobiliary disorders) | 0 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cholestatic icterus (Hepatobiliary disorders) | 0 | 0 | 1
Biliary fistula (Hepatobiliary disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No